CLINICAL TRIAL: NCT05698368
Title: A Digital Mindset Intervention to Improve Pain and Exercise Participation in Individuals With Knee Osteoarthritis: A Randomized, Parallel-group Study
Brief Title: Digital Knee Osteoarthritis Mindset Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Melissa Boswell, Study Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 69227
Record Dates: First submitted 2022-09-09; First posted 2023-01-26 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis
Keywords: Mindset; Physical Activity; Exercise; Psychology; Pain; Digital Health; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity; Pain; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three groups in parallel for the duration of the study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blind investigator and outcomes assessor: does not know group label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active comparator group (Active Comparator): A series of educational videos and reflective questions of the same duration and required attention as the mindset intervention program. The videos are sourced videos from YouTube that educate about osteoarthritis. The content consists of information about osteoarthritis that patients would typically receive if looking for more information about the disease, including disease pathology, risks, symptoms, and treatment strategies. The included videos contain factual content with a similar format to the mindset intervention videos, including live experts sharing information with animations and supplementary b-roll footage.
  Interventions: Other: Active comparator
- Mindset intervention group (Experimental): Four modules, each with a series of videos and reflective questions. Each module takes approximately 20-60 minutes to complete, with a total of about two hours to complete the entire program. Participants have one week to complete the program at their own pace. Participants are suggested to complete one module per day but are encouraged to go at the pace that works best for them.
  Interventions: Behavioral: Mindset intervention
- Waitlist control group (No Intervention): This group will take the same surveys as the other groups at the same time points but will not receive any additional content.

INTERVENTIONS:
Behavioral: Mindset intervention — Participants receive a digital mindset intervention to improve mindsets about osteoarthritis and exercise.
  Arms: Mindset intervention group
Other: Active comparator — Participants receive a series of osteoarthritis education videos and reflective questions that matches the digital mindset intervention in duration and attention.
  Other Names: Educational content
  Arms: Active comparator group

SUMMARY:
The aim of our clinical trial is to test if an online mindset intervention improves mindsets and physical activity levels more than an education intervention in individuals with knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis affects 7% of the global population and is a leading cause of disability globally. Physical activity improves health outcomes, weight management, and knee function for people with knee osteoarthritis and should be considered first-line treatment. Yet, physical activity levels in this population are low compared to those without knee osteoarthritis.

Existing knowledge: Emerging research has highlighted the powerful influence of mindsets about exercise on engagement in physical activity. Mindsets are core assumptions about a domain or category that orient individuals to a particular set of attributions, expectations, and goals (a "meaning system"). In individuals with knee osteoarthritis, mindsets about the appeal of physical activity relate to future physical activity levels and one's chosen symptom management strategy, and mindsets about osteoarthritis relate to knee symptoms.

The investigators developed a digital mindset intervention to improve mindsets about exercise and osteoarthritis in individuals with knee osteoarthritis. The investigators piloted the intervention on 21 individuals with knee osteoarthritis throughout the United States. Participants improved in exercise and osteoarthritis mindsets. However, this was a small sample size, a control group was not used, and it was cross-sectional, thus, not able to evaluate changes in physical activity and osteoarthritis symptoms.

Need for a trial: A digital, low-cost, and, thus, scalable intervention to improve mindsets about osteoarthritis and exercise may improve pain and function and physical activity levels for the millions of individuals affected with knee osteoarthritis. A large randomized trial is therefore needed to evaluate if our mindset intervention leads to improvements in physical activity levels and osteoarthritis symptoms and, further, if these changes are due to more adaptive mindsets about exercise and osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Over 45 years of age
* Self-reported doctor's diagnosis of knee osteoarthritis OR meets the National Institute for - - Health and Care Excellence osteoarthritis clinical criteria (activity-related knee pain and no knee morning stiffness lasting ≥ 30 minutes)
* Knee pain for at least 3 months
* Ability to walk unaided
* Can read and write in English
* Consistent internet access
* Willingness and ability to comply with the study requirements

Exclusion criteria:

* Past total knee arthroplasty or scheduled surgical procedure on any back or lower limb with osteoarthritis within the next 12 months
* Recent serious injury (within the past 2 months) on the knee(s) with osteoarthritis
* Any condition making it unsafe to participate in physical activity
* Intra-articular therapy within the past 6 months (e.g. injections such as corticosteroids and hyaluronic acid)
* Participates in physical exercise for 30 minutes or more 5 days per week

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Boswell, PhD, Principal Investigator — Stanford University; Scott Delp, PhD, Principal Investigator — Stanford University; Alia Crum, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data, including participant characteristics and outcome measures, will be made available after de-identification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon manuscript submission
Access Criteria: Open-source

REFERENCES:
- [Background] Boswell MA, Evans KM, Zion SR, Boles DZ, Hicks JL, Delp SL, Crum AJ. Mindset is associated with future physical activity and management strategies in individuals with knee osteoarthritis. Ann Phys Rehabil Med. 2022 Nov;65(6):101634. doi: 10.1016/j.rehab.2022.101634. Epub 2022 Apr 28. PMID 35091113
- [Background] Hinman RS, Campbell PK, Lawford BJ, Briggs AM, Gale J, Bills C, Kasza J, Harris A, French SD, Bunker SJ, Forbes A, Bennell KL. Does telephone-delivered exercise advice and support by physiotherapists improve pain and/or function in people with knee osteoarthritis? Telecare randomised controlled trial. Br J Sports Med. 2020 Jul;54(13):790-797. doi: 10.1136/bjsports-2019-101183. Epub 2019 Nov 20. PMID 31748198
- [Background] Crum AJ, Salovey P, Achor S. Rethinking stress: the role of mindsets in determining the stress response. J Pers Soc Psychol. 2013 Apr;104(4):716-33. doi: 10.1037/a0031201. Epub 2013 Feb 25. PMID 23437923
- [Background] Gay C, Guiguet-Auclair C, Mourgues C, Gerbaud L, Coudeyre E. Physical activity level and association with behavioral factors in knee osteoarthritis. Ann Phys Rehabil Med. 2019 Jan;62(1):14-20. doi: 10.1016/j.rehab.2018.09.005. Epub 2018 Oct 2. PMID 30290283
- [Background] Fransen M, McConnell S. Exercise for osteoarthritis of the knee. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD004376. doi: 10.1002/14651858.CD004376.pub2. PMID 18843657
- [Background] Marks R. Knee osteoarthritis and exercise adherence: a review. Curr Aging Sci. 2012 Feb;5(1):72-83. doi: 10.2174/1874609811205010072. PMID 21762086
- [Background] Hunter DJ, March L, Chew M. Osteoarthritis in 2020 and beyond: a Lancet Commission. Lancet. 2020 Nov 28;396(10264):1711-1712. doi: 10.1016/S0140-6736(20)32230-3. Epub 2020 Nov 4. No abstract available. PMID 33159851
- [Background] Stanton TR, Karran EL, Butler DS, Hull MJ, Schwetlik SN, Braithwaite FA, Jones HG, Moseley GL, Hill CL, Tomkins-Lane C, Maher C, Bennell K. A pain science education and walking program to increase physical activity in people with symptomatic knee osteoarthritis: a feasibility study. Pain Rep. 2020 Sep 24;5(5):e830. doi: 10.1097/PR9.0000000000000830. eCollection 2020 Sep-Oct. PMID 33490835
- [Background] Thorstensson CA, Garellick G, Rystedt H, Dahlberg LE. Better Management of Patients with Osteoarthritis: Development and Nationwide Implementation of an Evidence-Based Supported Osteoarthritis Self-Management Programme. Musculoskeletal Care. 2015 Jun;13(2):67-75. doi: 10.1002/msc.1085. Epub 2014 Oct 24. PMID 25345913
- [Background] Pisters MF, Veenhof C, Schellevis FG, De Bakker DH, Dekker J. Long-term effectiveness of exercise therapy in patients with osteoarthritis of the hip or knee: a randomized controlled trial comparing two different physical therapy interventions. Osteoarthritis Cartilage. 2010 Aug;18(8):1019-26. doi: 10.1016/j.joca.2010.05.008. Epub 2010 May 19. PMID 20488250
- [Background] Skou ST, Koes BW, Gronne DT, Young J, Roos EM. Comparison of three sets of clinical classification criteria for knee osteoarthritis: a cross-sectional study of 13,459 patients treated in primary care. Osteoarthritis Cartilage. 2020 Feb;28(2):167-172. doi: 10.1016/j.joca.2019.09.003. Epub 2019 Sep 17. PMID 31539621
- [Background] Boles DZ, DeSousa M, Turnwald BP, Horii RI, Duarte T, Zahrt OH, Markus HR, Crum AJ. Can Exercising and Eating Healthy Be Fun and Indulgent Instead of Boring and Depriving? Targeting Mindsets About the Process of Engaging in Healthy Behaviors. Front Psychol. 2021 Oct 5;12:745950. doi: 10.3389/fpsyg.2021.745950. eCollection 2021. PMID 34712186
- [Background] Washburn RA, Smith KW, Jette AM, Janney CA. The Physical Activity Scale for the Elderly (PASE): development and evaluation. J Clin Epidemiol. 1993 Feb;46(2):153-62. doi: 10.1016/0895-4356(93)90053-4. PMID 8437031
- [Background] Abbott JH, Hobbs C, Gwynne-Jones D; MOA Trial Team. The ShortMAC: Minimum Important Change of a Reduced Version of the Western Ontario and McMaster Universities Osteoarthritis Index. J Orthop Sports Phys Ther. 2018 Feb;48(2):81-86. doi: 10.2519/jospt.2018.7676. Epub 2017 Oct 21. PMID 29056072
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Darlow B, Abbott H, Bennell K, Briggs AM, Brown M, Clark J, Dean S, French S, Hinman RS, Krageloh C, Metcalf B, O'Brien D, Stanley J, Whittaker JL. Knowledge about osteoarthritis: Development of the Hip and Knee Osteoarthritis Knowledge Scales and protocol for testing their measurement properties. Osteoarthr Cartil Open. 2021 Apr 9;3(2):100160. doi: 10.1016/j.ocarto.2021.100160. eCollection 2021 Jun. PMID 36474995
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Shelby RA, Somers TJ, Keefe FJ, DeVellis BM, Patterson C, Renner JB, Jordan JM. Brief Fear of Movement Scale for osteoarthritis. Arthritis Care Res (Hoboken). 2012 Jun;64(6):862-71. doi: 10.1002/acr.21626. Epub 2012 Jan 30. PMID 22290689
- [Background] Lorig K, Chastain RL, Ung E, Shoor S, Holman HR. Development and evaluation of a scale to measure perceived self-efficacy in people with arthritis. Arthritis Rheum. 1989 Jan;32(1):37-44. doi: 10.1002/anr.1780320107. PMID 2912463
- [Derived] Boswell MA, Evans KM, Ghandwani D, Hastie T, Zion SR, Moya PL, Giori NJ, Hicks JL, Crum AJ, Delp SL. A randomized clinical trial testing digital mindset intervention for knee osteoarthritis pain and activity improvement. NPJ Digit Med. 2024 Oct 17;7(1):285. doi: 10.1038/s41746-024-01281-8. PMID 39414999

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator (Education) Group: A series of educational videos and reflective questions of the same duration and required attention as the mindset intervention program. The videos are sourced videos from YouTube that educate about osteoarthritis. The content consists of information about osteoarthritis that patients would typically receive if looking for more information about the disease, including disease pathology, risks, symptoms, and treatment strategies. The included videos contain factual content with a similar format to the mindset intervention videos, including live experts sharing information with animations and supplementary b-roll footage.
  Active comparator: Participants receive a series of osteoarthritis education videos and reflective questions that matches the digital mindset intervention in duration and attention.
- No-intervention (Survey-only) Control Group: This group will take the same surveys as the other groups at the same time points but will not receive any additional content.
Period: Overall Study
Arm/Group | Mindset Intervention Group | Active Comparator (Education) Group | No-intervention (Survey-only) Control Group
Started | 151 | 152 | 155
Completed | 130 | 135 | 143
Not Completed | 21 | 17 | 12

BASELINE CHARACTERISTICS:
Groups:
- Survey-only Group: This group will take the same surveys as the other groups at the same time points but will not receive any additional content.
- Total: Total of all reporting groups
Arm/Group | Active Comparator Group | Mindset Intervention Group | Survey-only Group | Total
Number analyzed (Participants) | 135 | 130 | 143 | 408
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (9.2) | 64.1 (8.0) | 63.0 (9.0) | 63.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 79 | 85 | 245
  Male | 54 | 51 | 58 | 163
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan NativeAmerican Indian or Alaskan Native | 4 | 2 | 3 | 9
  Asian | 7 | 7 | 2 | 16
  Black or African-American | 6 | 4 | 9 | 19
  Hispanic or Latino | 2 | 2 | 10 | 14
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0
  White | 118 | 118 | 128 | 364
  Other | 3 | 4 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Knee Pain Measured by Numeric Pain Rating Scale
Description: Knee pain scored from 0 - 10 (0 being no pain and 10 being the worst pain)
Time Frame: Change from Baseline at 1 month
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Comparator Group | Mindset Intervention Group | Survey-only Group
Number analyzed (Participants) | 135 | 130 | 143
units on a scale | -0.2 [-0.5 to 0.0] | -0.5 [-0.8 to -0.1] | -0.1 [-0.4 to 0.2]

2. Primary Outcome: Change From Baseline in Physical Activity Measured by Physical Activity Scale for the Elderly
Description: The Physical Activity Scale for the Elderly (PASE) asks respondents about the frequency of light, moderate, and strenuous work and leisure activities and is a validated measure of self-reported physical activity for individuals with osteoarthritis. The scale is scored from 0 (no physical activity) to 793 (very high physical activity).
Time Frame: Change from Baseline at 1 month
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Comparator Group | Mindset Intervention Group | Survey-only Group
Number analyzed (Participants) | 135 | 130 | 143
units on a scale | 32.6 [18.7 to 46.3] | 38.9 [24.3 to 53.6] | 10.3 [2.0 to 22.6]

3. Primary Outcome: Change From Baseline in Mindset About the Process of Health - Physical Activity (MPH-Physical Activity) Scale
Description: The Process of Health Mindset -- Exercise measure is a one-factor scale developed and validated to assess mindset about the process of engaging in physical activity (e.g., physical activity is difficult/easy, unpleasant/pleasurable, boring/fun). The scale consists of 7 items scored from 1 to 4, with a higher score reflecting a more appeal-focused mindset about physical activity, and then averaged for a total score between 1 to 4.
Time Frame: Change from Baseline at Post-intervention (immediately following intervention completion)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Comparator Group | Mindset Intervention Group | Survey-only Group
Number analyzed (Participants) | 135 | 130 | 143
units on a scale | 0.3 [0.2 to 0.3] | 0.5 [0.4 to 0.6] | 0.1 [0.0 to 0.1]

4. Primary Outcome: Change From Baseline in Osteoarthritis Mindset by the Illness Mindset Inventory
Description: The Illness Mindset Inventory measures three mindsets about the nature and meaning of illness: that it is a catastrophe, manageable, or an opportunity. The scale consists of 20 items measured on a 6-point scale and scored from 1 to 6, with 10 of those questions capturing mindsets about osteoarthritis. The extent to which a participant endorses a particular mindset can be obtained by calculating the mean score for each mindset. A higher score indicates greater agreement with the mindset. The investigators adapted the scale to focus on mindsets about "knee osteoarthritis" as opposed to "chronic disease." There are three subscales, Osteoarthritis is Castrophic, Osteoarthritis is Manageable, and Osteoarthritis is Opportunistic. The questions pertaining to each subscale are averaged for a total score from 1 to 6 for each subscale.
Time Frame: Change from Baseline at Post-intervention (immediately following intervention completion)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Comparator Group | Mindset Intervention Group | Survey-only Group
Number analyzed (Participants) | 135 | 130 | 143
units on a scale
  Osteoarthritis is Catastrophic | -0.5 [-0.6 to -0.3] | -1.1 [-1.3 to -1.0] | -0.2 [-0.3 to -0.1]
  Osteoarthritis is Manageable | 0.7 [0.5 to 0.8] | 1.1 [0.9 to 1.2] | 0.2 [0.1 to 0.3]
  Osteoarthritis is Opportunistic | 0.7 [0.6 to 0.8] | 1.1 [1.0 to 1.2] | 0.2 [0.0 to 0.3]

5. Secondary Outcome: Change From Baseline in Knee Pain and Functioning by the Short Version of Western Ontario and McMaster Universities Arthritis Index (shortMAC)
Description: The short-version of the Western Ontario and McMaster Universities Osteoarthritis Index (ShortMAC) is a disease-specific 12-item measure of knee pain, stiffness, and function. It has been validated and shown to be reliable in patients with knee osteoarthritis. It is measured on the Likert scale and can be divided into two subscales: pain and function. Pain subscore range, 0 (low pain) to 20 (high pain); Function subscore range, 0 (low difficulty) to 28 (high difficulty).
Time Frame: Change from Baseline at 1 month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Comparator Group | Mindset Intervention Group | Waitlist Control Group
Number analyzed (Participants) | 135 | 130 | 143
score on a scale
  Pain | -0.6 [-1.0 to -0.2] | -0.8 [-1.2 to -0.4] | -0.4 [-0.7 to 0.0]
  Function | -0.7 [-1.3 to -0.2] | -1.0 [-1.5 to -0.4] | -0.5 [-1.1 to 0.0]

6. Secondary Outcome: Change From Baseline in Knee Osteoarthritis Knowledge by the Knee Osteoarthritis Knowledge Scale
Description: The Knee Osteoarthritis Knowledge Scale is scored from 11-55 and measures knowledge about osteoarthritis in individuals with knee or hip osteoarthritis.
Time Frame: Change from Baseline at Post-intervention (immediately following intervention completion)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindset Intervention Group | Active Comparator (Education) Group | No-intervention (Survey-only) Control Group
Number analyzed (Participants) | 130 | 135 | 143
score on a scale | 10.5 [9.4 to 11.6] | 3.1 [2.2 to 4.0] | 0.6 [-0.1 to 1.4]

7. Secondary Outcome: Change From Baseline in Perceived Need for Surgery by a Surgery Perception Question
Description: Perceived need for surgery will be assessed by the single question, "How likely do you think you are of needing knee replacement surgery in the future?" It is answered on the Likert scale from 1 (very unlikely) to 5 (very likely). All items are averaged together for a final score between 1 to 5.
Time Frame: Change from Baseline at 1 month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindset Intervention Group | Active Comparator (Education) Group | No-intervention (Survey-only) Control Group
Number analyzed (Participants) | 130 | 135 | 143
score on a scale | -0.6 [-0.7 to -0.4] | -0.2 [-0.4 to 0.0] | 0.0 [-0.2 to 0.1]

8. Secondary Outcome: Change From Baseline in Symptom Management Strategy by an Osteoarthritis Symptom Management Question. The Variable is Reported as a % of Participants Who Reported Using the Symptom Management Strategy.
Description: Chosen symptom management strategy(ies) will be assessed by the single question, "Which of the following are ways in which you manage and/or improve your osteoarthritis symptoms? Please select all that apply." It is answer via multiple choice with multiple selection option. The options available are the most common strategies as determined by previous studies with an additional option for fill in. The reported value is the percentage of participants that selected the management strategy as a strategy they implement.
Time Frame: Change from Baseline at 1 month
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Mindset Intervention Group | Active Comparator (Education) Group | No-intervention (Survey-only) Control Group
Number analyzed (Participants) | 130 | 135 | 143
percentage
  Pain medications | -3.8 [-12.5 to 4.8] | 4.4 [-0.1 to 9.0] | -9.1 [-16.1 to -2.1]
  Injections | -6.2 [-13.8 to 1.5] | 3.7 [-4.1 to 11.5] | 0.7 [-5.9 to 7.3]
  Exercise | 20.8 [12.8 to 28.7] | 16.3 [7.2 to 25.3] | 6.3 [-1.5 to 14.1]
  Supervised physical therapy | -2.3 [-9.2 to 4.6] | 4.4 [-2.7 to 11.5] | -2.8 [-10.3 to 4.7]
  Rest | -1.5 [-10.7 to 7.0] | 11.1 [3.2 to 19.0] | -1.4 [-8.9 to 6.1]
  Imposing physical limitations | -19.2 [-28.3 to -10.1] | 5.2 [-4.3 to 14.7] | -7.7 [-16.8 to 1.4]
  Diet or weight management | 17.7 [8.2 to 27.0] | 14.8 [7.0 to 22.7] | 11.2 [3.1 to 19.2]
  Self-soothing | 10.0 [1.0 to 19.0] | 0.7 [-8.6 to 10.1] | -2.1 [-10.0 to 5.8]
  Mindset | 7.7 [-1.5 to 16.9] | -2.2 [-11.3 to 6.9] | -6.3 [-14.8 to 2.2]
  Nothing | 0.0 [-4.3 to 4.3] | -0.7 [-5.1 to 3.6] | -2.1 [-5.2 to 1.0]

9. Secondary Outcome: Change From Baseline in Fear of Movement by the Brief Fear of Movement Scale for Osteoarthritis
Description: The Brief Fear of Movement Scale for Osteoarthritis is a 6-item scale validated to assess fear of movement in individuals with osteoarthritis. All items are averaged for a final score range of 1 (low fear) to 4 (high fear).
Time Frame: Change from Baseline at 1 month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindset Intervention Group | Active Comparator (Education) Group | No-intervention (Survey-only) Control Group
Number analyzed (Participants) | 130 | 135 | 143
score on a scale | -0.4 [-0.5 to -0.3] | -0.2 [-0.7 to 0.5] | 0.0 [0.0 to 0.1]

10. Secondary Outcome: Change From Baseline in Arthritis Self-efficacy: Pain and Other Symptoms by the Arthritis Self-efficacy Pain and Other Symptoms Subscales
Description: The Arthritis-Self Efficacy Scale is scored from a 1 to 10 with higher scores indicating greater self-efficacy. The scale will be divided into the "pain" and "other symptoms" subscales. The items on each subscale are averaged for a final score from 1 to 10.
Time Frame: Change from Baseline at 1 month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindset Intervention Group | Active Comparator (Education) Group | No-intervention (Survey-only) Control Group
Number analyzed (Participants) | 130 | 135 | 143
score on a scale
  Pain | 1.4 [1.1 to 1.7] | 0.6 [0.4 to 0.9] | 0.1 [0.0 to 0.5]
  Other symptoms | 1.1 [0.9 to 1.4] | 0.6 [0.3 to 0.9] | 0.5 [0.3 to 0.8]

11. Secondary Outcome: Change From Baseline in Physical and Mental Health: Global Health: Patient-Reported Outcomes Measurement Information System (PROMIS) Scale v1.2 - Global Health (Physical and Mental Health Sub-scales)
Description: The PROMIS v.1.1 Global Health Short Form is a 10-item survey that measures overall physical function, fatigue, pain, emotional distress, and social health in healthy and clinical adult populations. It will be divided into two subscales: physical health and mental health. The Physical Health subscore ranges from 1 (poor) to 5 (excellent). The Mental Health subscore ranges from 1 (poor) to 5 (excellent).
Time Frame: Change from Baseline at 1 month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindset Intervention Group | Active Comparator (Education) Group | No-intervention (Survey-only) Control Group
Number analyzed (Participants) | 130 | 135 | 143
score on a scale
  Physical health | 0.2 [0.1 to 0.2] | 0.1 [0.0 to 0.2] | 0.0 [0.0 to 0.1]
  Mental health | 0.1 [0.0 to 0.2] | 0.0 [-0.5 to 0.5] | 0.0 [-0.1 to 0.06]

12. Secondary Outcome: Change From Baseline in Body Mindset by the Illness Mindset Inventory
Description: The Illness Mindset Inventory measures three mindsets about the nature of the body in the context of a chronic illness: that it is adversarial, responsive, or resilient. The scale consists of 20 items measured on a 6-point scale and scored from 1 to 6, with 10 of those questions capturing mindsets about the body. The extent to which a participant endorses a particular mindset can be obtained by calculating the mean score for each mindset. A higher score indicates greater agreement with the mindset. The investigators adapted the scale to focus on mindsets about "knee osteoarthritis" as opposed to "chronic disease." The three subscales are The Body is Adversarial, The Body is Capable, and the Body is Responsive. The items from each subscale are averaged for a final score between 1-6.
Time Frame: Change from Baseline at Post-intervention (immediately following intervention completion)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindset Intervention Group | Active Comparator (Education) Group | No-intervention (Survey-only) Control Group
Number analyzed (Participants) | 130 | 135 | 143
score on a scale
  The Body is Adversarial | -0.6 [-0.8 to -0.5] | -0.4 [-0.5 to -0.2] | -0.1 [-0.1 to 0.0]
  The Body is Capable | 1.3 [1.2 to 1.5] | 0.6 [0.4 to 0.7] | 0.2 [0.0 to 0.3]
  The Body is Responsive | 0.7 [0.5 to 0.8] | 0.4 [0.3 to 0.5] | 0.2 [0.0 to 0.2]

13. Secondary Outcome: Change From Baseline in Adequacy Mindset by the Adequacy of Activity Mindset Measure
Description: The Adequacy of Activity Mindset Measure is a scale developed to assess mindsets about the adequacy and benefits of ones' physical activity as it relates to health. The scale consists of 5 items measured on a 7-point scale and scored from 1 to 7, with a higher score reflecting a more adaptive mindset about the benefits and risks associated with current levels of physical activity. All items are averaged for a final score between 1 to 7.
Time Frame: Change from Baseline at Post-intervention (immediately following intervention completion)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindset Intervention Group | Active Comparator (Education) Group | No-intervention (Survey-only) Control Group
Number analyzed (Participants) | 130 | 135 | 143
score on a scale | 0.3 [0.1 to 0.5] | 0.2 [0.1 to 0.4] | 0.0 [-0.1 to 0.1]

ADVERSE EVENTS:
Time Frame: 5 months
Description: The definition did not differ. This study was low risk.
Arm/Group | Active Comparator Group | Mindset Intervention Group | Survey-Only Group
All-Cause Mortality (participants affected / at risk) | 0/135 | 0/130 | 0/143
Serious Adverse Events (participants affected / at risk) | 0/135 | 0/130 | 0/143
Other Adverse Events (participants affected / at risk) | 0/135 | 0/130 | 0/143

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT05698368/Prot_SAP_ICF_000.pdf